CLINICAL TRIAL: NCT01136226
Title: A 12 Month Open Label Study of Serum Testosterone Recovery and PSA After Neo-Adjuvant Treatment With Eligard(TM) 22.5mg Used With Radiation Therapy in Patients With Early Prostate Cancer
Brief Title: Evaluate Recovery of Testosterone for Patients Using Eligard
Acronym: Eligard
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chesapeake Urology Research Associates (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CURA-RT-001
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eligard (TM) (Other): Eligard (TM) administered 22.5mg
  Interventions: Drug: Eligard (TM)

INTERVENTIONS:
Drug: Eligard (TM) — Eligard (TM) 22.5 mg administered at baseline and Month 3

SUMMARY:
The purpose of this study is to determine if testosterone will recover to 90% by year 1 after using Eligard.

DETAILED DESCRIPTION:
This is a Multi-center, open-label study to evaluate testosterone recovery after six months of neo-adjuvant treatment with ELIGARD (TM) 22.5mg used with Radiation Therapy in patients with TNM T1, T2 or T3A adenocarcinoma of the prostate. The 60 patients will receive two subcutaneous administration of ELIGARD (TM) 22.5mg (Baseline and Month 3) and receive Radiation Therapy (Month 2-4).

ELIGIBILITY:
Inclusion Criteria:

* Must be outpatient, not hospitalized
* Male Patient between ages 50-80, inclusive
* Histologically/Cytologically graded adenocarcinoma of the prostate
* Must have T1, T2 or T3a adenocarcinoma of the prostate
* Must be a candidate for radiation therapy. Hormone refractory patients excluded
* WHO/ECOG score of 0,1 or 2

Exclusion Criteria:

* NO evidence of urinary tract that would put the patient at risk in the opinion of the Investigator.
* Used the following treatments for prostate Cancer

  *immunotherapy *chemotherapy *External Beam Radiation *brachytherapy *hormonal therapy *biological response modifiers
* Prior Prostate Surgery (excluding TUNA or TURP)
* Undergone Orchiectomy, adrenalectomy, hypophysectomy or be receiving any product which could alter the function of these organs
* Use of Investigational Drug, Biologic or device within five half-lives of its physiological action or three months prior to base line, whichever is longer
* Over the counter or alternative medical therapies which have estrogenic or anti-androgenic effect
* uncontrolled CHF within 6 months to baseline
* Myocardial Infarct, coronary vascular procedure or Clinically SignificantCardiovascualr Disease within 6 months of baseline Visit
* Venous thrombosis with in 6 Months of Screening
* Uncontrolled Hypertension defined as >170/100 or Symptomatic Hypotension within 3 months of Baseline
* Insulin dependant Diabetic Patients Must not administer in an anatomic region where they will receive Eligard.
* Drug or Alcohol Abuse 6 months prior to Baseline
* Other Serious Illness at the discretion of the Investigator
* Patients receiving anti-coagulant or anti-platlet medication must be on a stable dose for 3 months prior to Baseline
* Hypersensitivity to GnRH, GnRH agonists

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 2003-2008 at a medical office setting
Groups:
- Single Arm- Eligard: Eligard 22.5mg is only intervention administered
Period: Overall Study
Arm/Group | Single Arm- Eligard
Started | 42
Completed | 29
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm- Eligard
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone Recovery
Description: To Evaluate the time to testosterone recovery, which is defined as a return to with in 90% of pretreatment level, after 6 months of neo-adjuvant treatment with Eligard 22.5mg with Radiation Therapy in patients with early prostate Cancer
Time Frame: 6 mos
Measure: Mean (Full Range); unit: Months
Arm/Group | Single Arm- Eligard
Number analyzed (Participants) | 29
Months | 6 [1 to 18]

2. Secondary Outcome: Safety Assessments
Description: Assess frequency and severity of spontaneously reported AE's Changes between baseline and testosterone recovery in serum testosterone and pre biopsy PSA clinical evidence of Prostate cancer changes between baseline and testosterone recovery in health questionnaire
Time Frame: 6 months
Population: data were not collected
Arm/Group | Eligard (TM)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm- Eligard
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes